CLINICAL TRIAL: NCT06103162
Title: Comparison of Different Feeding Appliances for Cleft Palate Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amel Salem, Clinical professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #R-RP-7-23-2
Record Dates: First submitted 2023-10-15; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cleft Palate
Keywords: feeding appliance ,flexible, rigid
MeSH Terms: conditions — Cleft Palate; Muscle Rigidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 rigid feeding plate (Active Comparator): Heat cure polymerizing acrylic resin was used to fabricate the second appliance.
  Interventions: Device: flexible feeding plate
- group 2 flexible feeding plate (Active Comparator): One mm thick clear thermoplastic sheet was adapted over the cast using a vacuum-forming machine.
  Interventions: Device: flexible feeding plate
- special feeding appliance (Active Comparator): special feeding bottle
  Interventions: Device: flexible feeding plate

INTERVENTIONS:
Device: flexible feeding plate — One mm thick clear thermoplastic sheet was adapted over the cast using a vacuum-forming machine.
  Other Names: special feeding appliance

SUMMARY:
This study will compare flexible , rigid feeding plates and a special feeding bottle for children with cleft palate.

DETAILED DESCRIPTION:
This study will compare flexible , rigid feeding plates and a special feeding bottle for children with cleft palate.

The purpose of the present study will be explained to the patient's parents and informed consent will be obtained according to the guidelines on human research adopted by the Research Ethics Committee, Faculty of Dentistry, Tanta University.

ELIGIBILITY:
Inclusion Criteria:

* Infants with age range from 1-15 days.
* Unilateral cleft palate.
* Medically free subjects.
* Both males and females.

Exclusion Criteria:

* Patients older than 15 days.
* Syndromic patients with other defects in addition to cleft lip and palate.
* Patients with bilateral cleft lip and palate.
* Patients with previous presurgical infant orthopedic treatment.
* Medically compromised patients.-

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
The feeding efficiency | during 1 month
  The measure was defined as the volume of fluid transferred per unit time, in milliliters per minute (mL/min).

CONTACTS AND LOCATIONS:
Overall Officials: Amel AE salem, Principal Investigator — faculty of dentistry tanta university
Locations (1):
- faculty of dentistry Tanta University, Tanta, Egypt